CLINICAL TRIAL: NCT00655213
Title: Spontaneous Atrio Ventricular Conduction Preservation
Acronym: SAVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: J.M Davy - Principal investigator, CH Montpellier
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGXD02 - SAVER
Record Dates: First submitted 2008-04-01; First posted 2008-04-09 (Estimated); Last update posted 2008-04-09 (Estimated); Status verified 2008-04

CONDITIONS: Sinus Node Dysfunction; Bradycardia-Tachycardia Syndrome; Paroxysmal Atrioventricular Block
Keywords: Pacing, AV conduction disorders, minimized ventricular pacing, AF
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): AAISafeR mode programming
  Interventions: Device: Symphony D 2450; Device: Symphony DR 2550
- 2 (Active Comparator): DDD with long AV Delay programming
  Interventions: Device: Symphony D 2450; Device: Symphony DR 2550
- 3 (Active Comparator): DDDAMC mode programming
  Interventions: Device: Symphony D 2450; Device: Symphony DR 2550
- 4 (Other): AAISafer mode programming in non randomized patients
  Interventions: Device: Symphony D 2450; Device: Symphony DR 2550

INTERVENTIONS:
Device: Symphony D 2450
Device: Symphony DR 2550

SUMMARY:
In case of sinus node dysfunction, it is often necessary to choose the safer option provided by a DDD pacemaker even though the most appropriate mode of pacing is AAI mode.

In addition to saving energy, the latter mode allows spontaneous ventricular activation, the haemodynamic consequences of which are, in most cases, better than those obtained with dual chamber pacing.

Recent studies as the MOST study suggest also that ventricular desynchronization imposed by right ventricular apical pacing even when AV synchrony is preserved increases the risk of atrial fibrillation in patients with SND. Similar results were already given by anterior studies (PIPAF) which, taking into account the percentage of ventricular pacing, suggested that AF prevention algorithm in combination with a preserved native conduction are efficient in reducing AF burden.

However, current practice is to implant a dual chamber pacemaker to prevent the risk of atrioventricular block (AVB) even if DDDR pacing with a fixed long AV delay was found inefficient in reducing ventricular pacing and was associated with a high risk of arrhythmias.

The Symphony 2550 cardiac pacemaker offers pacing modes that automatically switch from AAI(R) mode to DDD(R) or DDI(R) in event of severe atrioventricular conduction disorder, irrespective of whether or not these are accompanied by an atrial arrhythmia, returning spontaneously to AAI(R) mode as soon as the spontaneous AV conduction has resumed. These 2 particular modes are called the AAI SafeR and DDD/AMC (R) mode.

The main differences between both modes are that (i) AAI SafeR does not trigger any AV Delay after a sensed or paced atrial event which allows long PR intervals or even limited ventricular pauses with no switch to DDD(R), while (ii) DDD/AMC (R) is able to optimize AV Delay after switching to DDD(R) according to measured spontaneous conduction times and to provide an acceleration in case of vaso-vagal syndrome. This pacing mode has previously been assessed in clinical studies.

This study intends to demonstrate that the automatic modes switching significantly reduce the percentage of ventricular pacing in patients implanted with a spontaneous AV conduction and reduce the occurrence of atrial arrhythmias, on a mid-term follow-up period, in comparison to standard DDD pacing with long AVDelay.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been primo-implanted with a Symphony™ 2550 or 2450 devices for less than 3 months
* Patient with a normal spontaneous AV conduction at rest (PR < 250 ms)
* Patient implanted for Sinus Node Dysfunction, Braycardia-Tachycardia Syndrome, carotid sinus syndrome/ vaso vagal syndrome or paroxistic AV Block
* Patient implanted with a bipolar right-atrial lead and ventricular lead available in the local market
* Patient has signed a consent form after having received the appropriate information

Exclusion Criteria:

* Permanent 1st, 2nd or 3rd AV block
* Patient having a medical status complying with one of the following cases
* patient suffering from sustained ventricular arrhythmias
* patient having sustained a myocardial infarction within the last month
* patient having undergone cardiac surgery within the last month
* patient suffering from severe aortic stenosis
* patient suffering from unstable angina pectoris
* patient presents with permanent atrial arrhythmias
* Patient is not able to understand the study objectives and protocol or refuses to co-operate
* Patient is not available for scheduled follow-up
* Patient has a life expectancy less than one year
* Patient is included into another clinical study
* Patient is minor or a pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
mean percentage of ventricular pacing between the randomized branches on a two-months period (M3 visit) | 2 months
mean percentage of ventricular pacing between the studied groups during the whole study (up to 1 year). | 12 months

SECONDARY OUTCOMES:
percentage of ventricular pacing two month after randomization versus the percentage reported at the end of the first month follow-up in AAIsafeR mode. | 12 months
AF burden relatively to the branch of the protocol | 12 months
evolution of conduction disturbances by documentings nature, number and duration of ario-ventricular blocks. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc DAVY, PhD, Principal Investigator — CH Montpellier
Locations (67):
- Belgium (7):
  - Onze lieve Vrouw ziekenhuis, Aalst
  - Clinique Louis Caty, Baudour
  - Hôpital universitaire Brugmann, Brussels
  - Europa ziekenhuis, Campus Saint Elisabeth Uccle
  - Heiling Hart van Jezus, Moen
  - Hôpital Vésale (univ.), Montigny-le-Tilleul
  - CHU - Tivoli, Tivoli
- France (19):
  - Centre Hospitalier, Aix-en-Provence
  - CH Albi, Albi
  - CHU d'Angers, Angers
  - CHU Jean Minjoz, Besançon
  - CH de CASTRES, Castres-mazamet
  - Hospice St-Jacques-Hôspital G.Montpied, Clermont-Ferrand
  - CHU - Hopital Michallon, Grenoble
  - CHRU de Lille - Hôpital Cardiologique, Lille
  - CHU de Limoges, Limoges
  - CH Montpellier, Montpellier
  - CH Emile Muller, Mulhouse
  - CHU de Nantes, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU de Nice, Nice
  - Clinique Bizet, Paris
  - CHU Pontchaillou, Rennes
  - CHU Hopital C. Nicolle, Rouen
  - InParys Cardiology, Saint-Cloud
  - CHU de Nancy, Vandœuvre-lès-Nancy
- Germany (23):
  - Marien Hospital, Bonn
  - Universitätskliniken Bonn, Bonn
  - St.Josef-Stift Bremen, Bremen
  - KH Holweide, Cologne
  - St. Salvator Krankenhaus Halberstadt, Halberstadt
  - Holzminden Praxis Bub, Holzminden
  - Hürth Sana, Hürth
  - Herzzentrum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum Lüdenscheid, Lüdenscheid
  - Städt. Kh. Lüneburg, Lüneburg
  - Univ. Mainz, Mainz
  - Univ. Marburg, Marburg
  - Klinkum Memmingen, Memmingen
  - Augustinum, München
  - Klinikum Bogenhausen, München
  - Rot-Kreuz Krankenhaus, München
  - Praxis Bitar, Peine
  - Uni Regensburg, Regensburg
  - Prof. Frey Praxis Starnberg, Starnberg
  - Uni Ulm, Ulm
  - Waren-Müritzklinikum, Waren
  - Klinikum Wolgast, Wolgast
- Italy (11):
  - Ospedale Moscati, Avellino
  - Ospedale Mellini, Chiari (BS)
  - Ospedale Civile, Conegliano (TV)
  - Ospedale S. G. Battista, Foligno (PG)
  - Ospedale Umberto I, Mestre (VE)
  - Ospedale Civile, Portogruaro (VE)
  - Istituto Policlinico, San Donato
  - Ospedale Civile, Sesto S. Giovanni (MI)
  - Ospedale Civile, Trento
  - Ospedale Civili Reuniti, Venezia
  - Ospedale Civile, Voghera
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Queens Hospital, Burton-on-Trent
  - Castle Hill Hospital, Hull
  - Leeds General Infirmary, Leeds
  - Barts and The London NHS Trust, London
  - St Thomas' Hospital,, London